CLINICAL TRIAL: NCT03205605
Title: Determination of Serum Oxybutynin Levels After Using Oxybutynin Transdermal Delivery System and Transdermal Gel With and Without Standardized Heat Application in Healthy Human Volunteers
Brief Title: Effect of Heat on Oxybutynin Release and Absorption From Oxybutynin Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP-00070850
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Heat Effect
MeSH Terms: interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- baseline patch (Other): patch
  Interventions: Drug: oxybutynin
- baseline gel (Other): gel
  Interventions: Drug: oxybutynin
- patch with heat (Other): patch
  Interventions: Drug: oxybutynin
- gel with occlusion (Other): gel
  Interventions: Drug: oxybutynin

INTERVENTIONS:
Drug: oxybutynin — patch
  Arms: baseline patch; patch with heat
Drug: oxybutynin — gel
  Arms: baseline gel; gel with occlusion

SUMMARY:
This research study is intended to determine the effect of heat and occlusion on oxybutynin products.

DETAILED DESCRIPTION:
This research study is intended to determine the effect of heat and occlusion on oxybutynin products. This study will use an oxybutynin patch and gel that have been approved by the Food and Drug Administration (FDA) and are already sold to customers in the United States; will not include any placebos.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, non-lactating women who are of any ethnic background between the age of 18 to 45 years old
2. Subjects must be non-smokers/tobacco users (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes) over the previous 2 months and are not currently using tobacco products
3. Provide written informed consent before initiation of any of the study procedures
4. Agree not to participate in another clinical trial/study or to participate in an investigational drug study for at least one month after the last study session
5. Able to adhere to the study restrictions and protocol schedule
6. Able to participate in all study sessions
7. Subjects have upper arms large enough to allow for placement of 200 cm2 [31 in2] area for applications of gel. The arm distance from the greater tubercle to the olecranon process should be a minimum of 30 cm. The circumference of the upper arms should be a minimum of 30 cm.
8. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination and medication history
9. Negative urine drug screening test (cannabinoids, amphetamines, barbiturates, benzodiazepine, cocaine, methadone, opiates, PCP)
10. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine transaminase (ALT) and aspartate aminotransferase (AST)
11. Have normal screening laboratories for urine protein and urine glucose
12. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each procedure day, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or a vasectomized partner
13. Agree not to donate blood to a blood bank throughout participation in the study and for at least three months after last procedure day
14. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
15. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-165 mmHg
    * Diastolic blood pressure 60-100 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion Criteria:

1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of any study session
2. Smokers/tobacco users (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patch or electronic cigarettes)
3. Participation in any ongoing investigational drug trial/study or clinical drug trial/study
4. History of chronic obstructive pulmonary disease or cor pulmonale, or substantially decreased respiratory reserve, hypoxia, hypercapnia or pre-existing respiratory depression
5. Active positive Hepatitis B, C and/or HIV serologies
6. Positive urine drug screening test
7. Use of chronic prescription medications during the period 0 to 30 days; or over-the-counter medication (e.g. bisphosphonates [to treat osteoporosis], anticholinergics [used to treat diseases like asthma, incontinence, gastrointestinal cramps, and muscular spasms], antihistamines, topical corticosteroids) and short term (<30 days) prescription medications during the period 0-3 days before a study session [vitamin, herbal supplements and birth control medications not included)]
8. Donation or loss of greater than one pint of blood within 60 days of entry to the study
9. Any prior allergies to oxybutynin, other ingredients in the patch, gel or oral tablet tested, to medical tape products or other skin patches
10. Subject has problems with urinary retention, gastric retention or gastrointestinal obstruction
11. Subject has ulcerative colitis
12. Subject has gastric reflux disease or esophagitis
13. Subject has uncontrolled narrow-angle glaucoma
14. Subject has myasthenia gravis
15. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within one month before enrollment in this study or expects to receive an experimental agent during the study
16. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
17. Consumption (food or drink) of alcohol within 24 h prior to dose administration
18. History as either reported by the subject or evident to the investigator of infectious disease or skin infection or of chronic skin disease (e.g., psoriasis, atopic dermatitis)
19. History of diabetes
20. Hereditary skin disorders or any skin inflammatory conditions as reported by the volunteer or evident to the MAI
21. History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites
22. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site (upper arms), sunburn, raised moles and scars, open sores at application site (upper arms), scar tissue, tattoo, or coloration that would interfere with placement of products, skin assessment, or reactions to oxybutynin
23. BMI ≥30 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra L Stinchcomb, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy; Hazem E Hassan, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy
Locations (1):
- General Clinical Research Center (GCRC) at the University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin Patch and Gel: First study session received one oxybutynin patch (Oxytrol for Women), then at least one week washout period Second study session received oxybutynin gel (Gelnique), then at least one week washout period Third study session received one oxybutynin patch (Oxytrol for Women) with early and late heat (90 minutes) exposure, then at least one week washout period Fourth study session received oxybutynin gel (Gelnique) with occlusion (3 hours)
Period: Overall Study
Arm/Group | Oxybutynin Patch and Gel
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxybutynin Patch and Gel
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.08 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: PK Parameter
Description: Cmax (oxybutynin) during first heat period for patch (24-25.5 h)
Time Frame: 24 h, 24 h 15 min, 24 h 30 min, 24 h 45 min, 25 h, 25 h 15 min, 25 h 30 min post patch application
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Oxytrol for Women Patch (Baseline): baseline (no heat exposure)
- Oxytrol for Women Patch (Heat Exposure): external heat exposure at 24-25.5 h and 30-31.5 h
Arm/Group | Oxytrol for Women Patch (Baseline) | Oxytrol for Women Patch (Heat Exposure)
Number analyzed (Participants) | 13 | 12
ng/mL | 3.38 (0.63) | 30.75 (20.31)

2. Primary Outcome: PK Parameter
Description: Serum concentration (oxybutynin) at 30 h time point (patch removal)
Time Frame: 30 h post patch application
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Oxytrol for Women Patch (Baseline) | Oxytrol for Women Patch (Heat Exposure)
Number analyzed (Participants) | 13 | 12
ng/mL | 4.06 (1.24) | 12.99 (10.02)

3. Primary Outcome: PK Parameter
Description: Cmax (oxybutynin) at second heat exposure (30-31.5 h); after patch removed
Time Frame: 30 h, 30 h 15 min, 30 h 30 min (patch removed at 30 h)
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Oxytrol for Women Patch (Baseline) | Oxytrol for Women Patch (Heat Exposure)
Number analyzed (Participants) | 13 | 12
ng/mL | 4.96 (1.19) | 22.43 (15.14)

4. Primary Outcome: PK Parameter
Description: Cmax (oxybutynin)
Time Frame: 0 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 7 h 15 min, 7 h 30 min, 7 h 45 min, 8 h, 8 h 15 min, 8 h 30 min, 8 h 45 min, 9 h, 9 h 15 min, 9 h 30 min, 9 h 45 min, 10 h, 10 h 30 min, 11 h, 11 h 30 min, 12 h post gel application
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Gelnique Gel (Baseline): Gelnique gel applied for 12 h duration; no occlusion
- Gelnique Gel (Occlusion): Gelnique gel applied for 12 h duration; occluded from 7-10 h
Arm/Group | Gelnique Gel (Baseline) | Gelnique Gel (Occlusion)
Number analyzed (Participants) | 12 | 12
ng/mL | 5.00 (2.09) | 71.93 (32.21)

5. Primary Outcome: PK Parameter
Description: Cmax (N-desethyl oxybutynin)
Time Frame: as for outcome 4
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Gelnique Gel (Baseline) | Gelnique Gel (Occlusion)
Number analyzed (Participants) | 12 | 12
ng/mL | 0.36 (0.09) | 2.38 (0.62)

ADVERSE EVENTS:
Time Frame: For Study Session 1 & 3, 34 h 30 min post initial patch application followed by up to 72 h phone follow up. For Study Session 2 & 4, 12 h during gel application followed by up to 72 h phone follow up. If there was an adverse event, volunteers were followed up until adverse event resolved.
Arm/Group | Baseline Patch | Baseline Gel | Patch With Heat | Gel With Occlusion
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 7/13 | 10/12 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Patch (N=13) | Baseline Gel (N=13) | Patch With Heat (N=12) | Gel With Occlusion (N=12)
Pain at IV site (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
vesicle (blister) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Decreased blood pressure (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
ERYTHEMA (skin reddening) (Skin and subcutaneous tissue disorders) | 11 (11) | 7 (7) | 10 (10) | 10 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT03205605/Prot_SAP_000.pdf